CLINICAL TRIAL: NCT04583462
Title: Impact of Metformin on Peripheral Arterial Calcification in Type 1 Diabetes: a Double Blind Randomized Controlled Trial
Brief Title: Impact of Metformin on Peripheral Arterial Calcification in Type 1 Diabetes
Acronym: IMPACT-1D
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D20180102; 2018-003121-29 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes; Peripheral Arterial Calcification
Keywords: Metformin; Peripheral arterial calcification; Type 1 diabetes; Placebo
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin, started at 500 mg per day per os and titrated up to 2000 mg during 2 years (increase of 500 mg every two weeks)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo (coated tablet similar to metformin tablet titrated following the same schedule as in the experimental arm), started at 500 mg per day per os and titrated up to 2000 mg during 2 years (increase of 500 mg every two weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin, started at 500 mg per day per os and titrated up to 2000 mg during 2 years (increase of 500 mg every two weeks)
  Other Names: Metformine Arrow LAB 1000 mg
  Arms: Metformin
Drug: Placebo — Control group : Placebo (coated tablet similar to metformin tablet titrated following the same schedule as in the experimental arm) started at 500 mg per day per os and titrated up to 2000 mg during 2 years (increase of 500 mg every two weeks)
  Other Names: Control group
  Arms: Placebo

SUMMARY:
Vascular calcification (VC) is a complication frequently observed in elderly, in chronic kidney disease (CKD) and in diabetes (particularly in type 1 diabetes). VC is a dynamic pathophysiological process that causes cardiovascular morbidity and is an independent risk factor of major amputation. In vitro and human observational studies have suggested a role of metformin in preventing VC. The investigators propose to test the effect of metformin treatment during two years on lower limb arterial calcification evaluated by CT-scan in patients with type 1 diabetes and without CKD.

This research is a phase III double blind randomized controlled trial consisting of 2 years double-blind treatment phase (patients randomized to metformin or placebo) in type 1 diabetic patients.

The participants and the investigators will be blinded to the study medications taken during the double-blind treatment period

DETAILED DESCRIPTION:
The main objective of this study is to show that metformin, in patients with type 1 diabetes but without chronic kidney disease, is able to slow below- knee arterial calcification evaluated by the difference between below-knee arterial calcification score evaluated by CT-scan at T0 and T2years in type 1 diabetic patients treated or not with metformin. This research is a phase III double blind randomized controlled trial consisting of 2 years treatment phase (patients randomized to metformin or placebo).The participants and the investigators will be blinded to the study medications taken during the treatment period. The treatment delivered will be metformin vs placebo started at 500 mg per day per os and titrated up to 2000 mg (increase of 500 mg every two weeks). The duration of the treatment will be two years. The main inclusion criteria are: Type 1 diabetes / Women and Men ≥ 18 years old and ≤ 80 years old with complications: diabetic retinopathy and/or nephropathy (with creatinine clearance ≥ 60 mL/mn) and/or neuropathy and/or peripheral arterial occlusive disease and/or cardiopathy and/or stroke and/or cardiovascular risk factors (hypertension and/or dyslipidemia (HDL < 0.35g/L or LDL > 1.9g/L or treated dyslipidemia) and/or tobacco use (old or active smoking greater than 5 pack years))and/or Diabetes duration >20 years.

The secondary objectives and endpoints are: 1. To show that metformin, in patients with type 1 diabetes but without CKD, is able to slow below-knee arterial occlusive disease evaluated by the difference between below-knee arterial ultrasonographic occlusion score at T0 and T2years in type 1 diabetic patients supplemented or not with metformin, 2. To show that metformin, in patients with type 1 diabetes but without CKD, is able to improve ankle and toe brachial indexes evaluated by the difference between ankle and toe brachial indexes at T0 and T2years in type 1 diabetic patients supplemented or not with metformin, 3. To show that metformin, in patients with type 1 diabetes but without CKD, is able to improve pulse wave velocity evaluated by the difference between pulse wave velocity at T0 and T2 years in type 1 diabetic patients supplemented or not with metformin, 4. To show that metformin, in patients with type 1 diabetes but without chronic kidney disease, is able to slow coronary arterial calcification evaluated by the difference between coronary calcification score evaluated by CT-scan at T0 and T2years in type 1 diabetic patients treated or not with metformin, 5. To conduct a subgroup analysis for the primary outcome to evaluate whether the effect of metformin on the difference of below-knee arterial calcification score evaluated by CT-scan at T0 and T2years varies according to initial below-knee arterial calcification score (≤ versus >400) evaluated by the difference between below-knee arterial calcification score progression between T0 and T2years in type 1 diabetic patients treated or not with metformin and with initial below-knee arterial calcification score ≤ and >400.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes
2. Women and Men ≥ 18 years old and ≤ 80 years old with:

   * Complications: diabetic retinopathy and/or nephropathy (with creatinine clearance ≥ 60 mL/mn) and/or neuropathy and/or peripheral arterial occlusive disease and/or cardiopathy and/or stroke and/or
   * cardiovascular risk factors : hypertension and/or dyslipidemia (HDL < 0.35g/L or LDL > 1.9g/L or treated dyslipidemia) and/or tobacco use (old or active smoking greater than 5 pack years) and/or
   * Diabetes duration >20 years
3. For women in childbearing age, effective contraception during the whole trial
4. Signed written informed consent
5. Affiliation of a social security regime (AME excluded)

Exclusion Criteria:

1. Creatinine clearance of less than 3 months <60 mL/mn (MDRD) at the inclusion time
2. Known metformin contra-indication: severe liver insufficiency -CHILD B or C, heart failure (FEVG<45%) or history of pulmonary edema, respiratory insufficiency with history of acute respiratory failure or patients receiving oxygen therapy, chronic ethylism, lactic acidosis
3. Know sensitivity to metformin or to any of its excipients or placebo excipients (lactose)
4. Indication or history of lower limb angioplasty (with stenting) and/or bypass
5. Previous treatment with metformin (within 3 months prior to inclusion)
6. HbA1c of less than 3 months >11%
7. Chronic inflammatory disease or chronic immune-suppressive drugs intake
8. Participation in an another interventional trial (Jardé 1 and 2) or in the exclusion period of any other interventional study
9. Pregnancy woman (confirmed by a sanguine beta-human chorionic gonadotropin test) or breastfeeding woman
10. Patient under legal protection measure (tutorship or curatorship) or deprived of freedom
11. Unable to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Change between below-knee arterial calcification score evaluated by CT-scan at T0 and T2years in type 1 diabetic patients treated or not with metformin. | Change between T0 baseline visit and T2 years
  Below-knee artery calcification scores will be obtained after scanning with a 128-slice multidetector CT scanner without contrast, in a craniocaudal direction, from the bottom of the patella down to the ankle region. The 3-mm cross-sectional slices were separately analyzed. Analysis was performed by radiologists kept blind about the results of the color duplex ultrasonography, laboratory tests, and clinical examinations, using a commercially available software package (Heartbeat CaScore; Philips Healthcare). On cross-sectional images, areas of calcification along below-knee arteries with a density ≥130 Hounsfield units attenuation and a surface >1 mm2 were identified automatically. Calcification score, determined according to the method described by Agatston et al, will be obtained separately for each of the main below-knee arteries (distal popliteal, anterior tibial, posterior tibial, and peroneal arteries) and added up to obtain the calc

SECONDARY OUTCOMES:
Change between below-knee arterial ultrasonographic occlusion score at T0 and T2years in type 1 diabetic patients treated or not with metformin. | Change between T0 baseline visit and T2 years
  Detailed colour duplex ultrasonography will be performed, from the abdominal tree down to the foot arteries, to all the patients, by one physician by center. Occlusive disease will be defined as the presence of either >70% stenosis or an occlusion in any artery being studied (aorto-ilio-femoral segment, popliteal artery, tibio-peroneal trunk, anterior tibial, posterior tibial, peroneal, and dorsalis pedis arteries). The results will be scored according to an adapted version of an angiographic score based on the severity of the stenosis in the lower limb arteries: 0 if stenosis is <70%, 2 if stenosis is >70%, and 3 in case of occlusion. Consequently, duplex scores range from 0 to 39. Mediacalcosis will be also graded for each infrapopliteal artery (popliteal arteries included): 0 if not visible, 1 if mild and discontinuous, 2 if continuous, and 3 if severe with lumen obstruction. Therefore, mediacalcosis scores range from 0 to 36.
Change between ankle and toe brachial indexes at T0 and T2years in type 1 diabetic patients supplemented or not with metformin. | Change between T0 baseline visit and T2 years
  Dorsalis pedis, posterior tibial and brachial arterial systolic blood pressures were measured with a Doppler probe (Parks Medical Electronics, Aloha, OR, USA). Measurements will be taken after participants have rested for 10 min in the supine position. Brachial blood pressure will be measured in the dominant arm with an appropriately sized cuff after 10 min rest in the supine position. Two measurements will be obtained and averaged.
  Toe systolic pressure measurements will be taken with the Systole Automated Toe Pressure System (Atys Medical, Soucieu-en-Jarrest, France)
Change between pulse wave velocity at T0 and T2years in type 1 diabetic patients supplemented or not with metformin. | Change between T0 baseline visit and T2 years
  Pulse Wave Velocity and pulse wave analysis were measured with applanation tonometry, using SphygmoCor system version 7.1 (Atcor Medical). Central arterial pressure (CAP) and central systolic pressure were derived and central augmentation index (AIx) was calculated. As AIx is influenced by heart rate, an index normalized for a heart rate of 75 beats/min was used. To determine pulse wave velocity, pulse wave forms were recorded at the right carotid artery and left femoral artery sequentially. Wave-transit time was calculated using the R-wave of a simultaneously recorded electrocardiogram as a reference frame.
Change between coronary calcification score evaluated by CT-scan at T0 and T2years in type 1 diabetic patients treated or not with metformin. | Change between T0 baseline visit and T2 years
  Agatston score is a semi-automated tool to calculate a score based on the extent of coronary artery calcification detected by an unenhanced low-dose CT scan, which is routinely performed in patients undergoing cardiac CT. Coronary artery calcification scores will be obtained after scanning with a 128-slice multidetector CT scanner without contrast, in a craniocaudal direction. Analysis was performed by radiologists kept blind about the results of laboratory tests and clinical examinations, using a commercially available software package (Heartbeat CaScore; Philips Healthcare). On cross-sectional images, areas of calcification along coronary arteries with a density ≥130 Hounsfield units attenuation and a surface >1 mm2 were identified automatically. Calcification score, determined according to the method described by Agatston et al, will be obtained separately for each of the main coronary arteries and added up to obtain the total coronary
Change between below- knee arterial calcification score progression between T0 and T2years with initial below-knee arterial calcification score ≤ and >400 (subgroup analysis) | Change between T0 baseline visit and T2 years
  Detailed colour duplex ultrasonography will be performed, from the abdominal tree down to the foot arteries, to all the patients, by one physician by center. Occlusive disease will be defined as the presence of either >70% stenosis or an occlusion in any artery being studied (aorto-ilio-femoral segment, popliteal artery, tibio-peroneal trunk, anterior tibial, posterior tibial, peroneal, and dorsalis pedis arteries). The results will be scored according to an adapted version of an angiographic score based on the severity of the stenosis in the lower limb arteries: 0 if stenosis is <70%, 2 if stenosis is >70%, and 3 in case of occlusion. Consequently, duplex scores range from 0 to 39. Mediacalcosis will be also graded for each infrapopliteal artery (popliteal arteries included): 0 if not visible, 1 if mild and discontinuous, 2 if continuous, and 3 if severe with lumen obstruction. Therefore, mediacalcosis scores range from 0 to 36.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier OB Bourron, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpêtrière Hospital, AP-HP, Diabetology department, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, National Commission for Information Technology and Freedoms) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.